CLINICAL TRIAL: NCT06601023
Title: Problem Management Plus Mindfulness-informed LegalEducation (PM+MiLE) for Addressing Gender-based Violence and Improving Parenting in Nigeria: a Randomised Control Trial
Brief Title: Problem Management Plus Mindfulness-informed Legal Education for Addressing Gender-based Violence and Improving Parenting
Acronym: PM+MiLE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Teesside University (Other)
Collaborators: Jos University Teaching Hospital (Other); University of Manchester (Other)
Responsible Party: Principal Investigator, Tarela Ike, Senior Lecturer and Principal Investigator, Teesside University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0000-0003-0516-0313e; PM+MiLE (Other: Teesside University)
Record Dates: First submitted 2024-09-14; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Depression, Anxiety; Trauma; Anxiety; Parenting Intervention; Woman Abuse; Child Behaviour; Stress
Keywords: Depression; Stress; Anxiety; Trauma; Gender-based violence; Parenting; Domestic violence; Women
MeSH Terms: conditions — Depression; Anxiety Disorders; Wounds and Injuries | interventions — Psychosocial Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Problem Management plus Mindfulness-informed LegalEducation (PM+MiLE) (Experimental): The PM+MiLE is a six sessions intervention lasting approximately 90 minutes. A session will be delivered weekly for six week.
  Interventions: Behavioral: Psychosocial intervention
- Control - Waitlist Group (No Intervention): The control group will receive no intervention until after the assessment periods at baseline, end of intervention and 3 months follow up before they will be administered the PM+MiLE.

INTERVENTIONS:
Behavioral: Psychosocial intervention — The PM+MiLE is a low-intensity intervention. The intervention will cover relevant aspects of brief mindfulness, legal education, awareness of human rights and challenges of complaint, including support. The problem management ambit will include understanding adversity, managing stress, managing problems, getting going and keep doing, strengthening social support and staying well and looking forward, including positive behaviour modification.The intervention will also incorporate child development and building positive parenting interactions with children.
  Arms: Problem Management plus Mindfulness-informed LegalEducation (PM+MiLE)

SUMMARY:
Gender-based violence and, more specifically, domestic violence is a prevalent problem globally and in Nigeria. Its effect significantly impacts women and also the wellbeing of their families. Limited access to support has posed a constraint in effectively addressing the issues suffered by affected victims in Nigeria. In addition, gender-based violence could affect parenting due to factors such as anxiety, trauma, depression, poor social support, limited awareness of legal channels for complaint and harsh parenting to children. The implication is that it could not only have a negative impact on the affected victim but also on their parenting styles or caring responsibilities, which could be detrimental to the child development, wellbeing and the potential subsequent resort to criminal behaviours. In essence, the current study aims to test the feasibility and acceptability of a novel cross disciplinary intervention titled, Problem Management plus Mindfulness-informed Legal Education (PM+MiLE) for addressing gender-based violence and improving parenting in Nigeria in comparison to the waitlist control group for the purposes of improving social cohesion, legal awareness, wellbeing and reducing depression, including trauma and anxiety as a result of experiencing gender-based violence, in Nigeria.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above
* Female with child(ren) or with caring responsibilities for child(ren).
* Able to provide full consent for their participation.
* A resident of the study areas (Delta, Jos, Lagos State, etc.)

Exclusion Criteria:

* Less than 18 years
* Unable to consent
* Currently undergoing severe mental healthtreatment
* Unable to speak the English language fl uently

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-09-24 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Service Satisfaction Scale | 6 weeks at the end of intervention
  A five item scale that can be used to assess and measure satisfaction, acceptability and quality of the intervention. Higher score denote positive outcomes and acceptability. Lower score denotes poor satisfaction and acceptability.

SECONDARY OUTCOMES:
Gender-based Violence, Stress and Parenting Scale | Baseline, end of intervention and 3 months post intervention.
  The scale is a 4 item scale that will be use for assessing and measuring gender-based violence, stress and parenting. The scale has an overall rating of 20 with score ranging 1-5 indicating severe stress in parenting, 5-10 indicating moderately severe stress in parenting, 11-15 mild stress in parenting and 16- 20 no stress in parenting.
Post-traumatic Stress Disorder Checklist (PCL-5) | Baseline, 6 weeks end of intervention and 3 months post intervention.
  The PCL-5 is a 20-item self-report measure that can be used to assess the 20 DSM-5 symptoms of post traumatic stress disorder. A 5-10 point change represents reliable change (i.e., change not due to chance) and a 10-20 point change represents clinically significant change.
Generalised Anxiety Disorder (GAD-7) | Baseline, 6 weeks end of intervention and 3 months post intervention.
  The GAD-7 is a seven item scale for screening, measuring and assessing the severity of generalised anxiety disorder.
  Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
Oslo Social Support Scale (OSSS-3) | Baseline, 6 weeks end of intervention and 3 months post intervention.
  The scale is a 3-item self-reported measure designed for assessing and measuring the level of social support.
  The sum score ranges from 3 to 14, with high values representing strong levels and low values representing poor levels of social support as indicated as follows: a) 3-8 poor social support, b) 9-11 moderate social support, c) 12-14 strong social support.
Legal-informed Awareness of Complaint Channel Scale (LACCS) | Baseline, 6 weeks end of intervention and 3 months post intervention.
  The LACCS is a 10-item scale that is designed for assessing and measuring level of awareness of complaint channels and legal rights. The scale has an overall rating of 30, with 0-7 indicating poor knowledge, 8-15 (average knowledge), 16-22 (good knowledge) and 23-30 (excellent knowledge).
Harsh Parenting Scale | Baseline, 6 weeks end of intervention and 3 months post intervention.
  The scale is a 4 item scale use to assess harsh parenting. The scale has a rating of 20 with lower scores indicating non harsh parenting and higher scores indicating severe harsh parenting.
Parenting Stress Scale | Baseline, 6 weeks end of intervention and 3 months post intervention.
  The PSS is an 18-item questionnaire for assessing parents' feelings about their parenting role, exploring both positive aspects (e.g. personal development, emotional benefits,) and negative aspects of parenthood (e.g. demands on resources, and feelings of stress). Parental stress scores range from 18 to 90, with lower scores indicating lower levels of parental stress.
European Quality of Life Scale EQ-5D-5L | Baseline, 6 weeks end of intervention and 3 months post intervention.
  The EQ-5D-5L is a 5 item scale designed to aid assessment of the generic quality of life.
  In the EQ-5D-5L, each dimension has five response levels: no problems (Level 1); slight (Level 2); moderate (Level 3); severe (Level 4); and extreme problems (Level 5). There are 3,125 possible health states defined by combining one level from each dimension, ranging from 11111 (full health) to 55555 (worst health).
Patient Health Questionnaire (PHQ-9) | Baseline, 6 weeks end of intervention and 3 months post intervention.
  This The Patient Health Questionnaire (PHQ-9) is a 9-item questionnaire that will be used for screening, monitoring, measuring and assessing the severity of depression.
  Low scores (e.g. 0-4) indicate no depression, however, higher scores (20-27) indicates severe depression.

IPD SHARING:
Plan to Share IPD: No
Data supporting this study cannot be made available due to the sensitive nature and ethical reasons on confidentiality.

REFERENCES:
- [Background] Oladepo O, Yusuf OB, Arulogun OS. Factors influencing gender based violence among men and women in selected states in Nigeria. Afr J Reprod Health. 2011 Dec;15(4):78-86. PMID 22571109
- [Background] Aborisade, R.A., (2024). Violence In A Patriarchal Nigerian Society. Routledge International Handbook of Investigative Interviewing and Interrogation, p.372.